CLINICAL TRIAL: NCT04591743
Title: Effectiveness of Transcranial Magnetic Stimulation (TMS) in Smoking Cessation, Combining Withdrawal Stimulation Followed by Maintenance Stimulation to Prevent Relapse: Single-center, Randomized, Controlled, Blinded Pilot Study
Brief Title: Effectiveness of Transcranial Magnetic Stimulation (TMS) in Smoking Cessation, Combining Withdrawal Stimulation Followed by Maintenance Stimulation to Prevent Relapse.
Acronym: TabacStim2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TROJAK CRBFC-E 2019
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Device: Active TCS; Drug: nicotine treatment; Other: Questionnaires
- Placebo group (Placebo Comparator)
  Interventions: Device: Placebo TCS; Drug: nicotine treatment; Other: Questionnaires

INTERVENTIONS:
Device: Active TCS — TCS active at 1 Hz on the right DLPFC for 6 weeks
  Arms: Experimental group
Device: Placebo TCS — Inactive TCS (placebo coil) at 1 Hz on right DLPFC for 6 weeks
  Arms: Placebo group
Drug: nicotine treatment — at least 21/14/7 mg/d + oral nicotine cp from 2 to 30 mg/d)
Other: Questionnaires — EVA on "craving", TCQ, QSU, BDI-II, CO tester, IGT, BART

SUMMARY:
Tobacco control is a Public Health priority. Tobacco is directly responsible for 75,000 deaths per year in France. Without help, less than 5% of smokers are still abstinent within 12 months of quitting. The use of nicotine substitutes only increases the chances of success in smoking cessation by 2 to 3%.

Brain imaging research shows that the dorsolateral prefrontal cortex (DLPFC) is involved in tobacco addiction. Disorders induced in the CPFDL cause an irrepressible desire to smoke (craving) and explain a large part of the relapse at the time of smoking cessation.

Transcranial magnetic stimulation (TMS) could be promising in smoking cessation. This technique allows direct stimulation of the DLPFC via a magnetic coil, so as to reduce the cortical activity of the DLPFC, and thus reduce tobacco craving.

A first randomized controlled study was conducted at the Dijon University Hospital in Dijon in smokers who were heavily addicted and who had failed with the usual withdrawal strategies. In this study, it was found that the combination of nicotine substitutes (to reduce the physical symptoms of withdrawal) with 10 sessions of TCS (to reduce craving) made it possible to maintain abstinence from tobacco during the first 2 weeks of withdrawal (% abstinence = 88.8% active TCS group vs. 50% placebo TCS group; p=0.027).

However, in this study, the therapeutic effect of the nicotine-TCS combination was not prolonged once the stimuli stopped. At 6 and 12 weeks from the start of withdrawal, abstinence rates in the active SMT and placebo SMT groups were no longer significantly different.

It is therefore proposed to renew the protocol by adding maintenance brain stimulation to the initial protocol. Used in the treatment of depression, the maintenance brain stimuli could increase the chances of smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has given oral consent
* Adult patient
* Patient wishing to stop smoking
* Patient highly addicted to nicotine (≥ score 7 on Fagerström's self-questionnaire*)
* Patient with at least 1 previous smoking cessation failure using recommended drug therapies (nicotine, vareniciline, bupropion)

Exclusion Criteria:

* Patient not affiliated or not benefiting from national health insurance
* Person deprived of their liberty by judicial or administrative decision
* Protected adults (curatorship, guardianship)
* Pregnant, parturient or breastfeeding woman
* Patient of childbearing age with a positive pregnancy test at inclusion
* Major patient incapable or unable to express consent
* Patient abstinent in the previous 3 months
* Patient with a substance use disorder (DSM-5 criteria) with other psychoactive substances other than tobacco
* Patient with a contraindication to the practice of TCS; personal history of seizure, pacemaker, neurosurgical clips, carotid or aortic clips, heart valves, hearing aid, ventricular bypass valve, sutures with wires or staples, foreign bodies in the eye, shrapnel, other prosthesis or cephalic ferromagnetic material.
* Patient employed by the investigator or trial site
* Patient with severe depression, defined by a score greater than or equal to 24 on the Hamilton Depression Rating Scale
* Patient who has had a recent change (< 1 month) in the prescription of psychotropic treatment
* Patient with severe and/or chronic psychiatric disorders, including schizophrenia, paranoia, and bipolar disorders type I and II.
* Patient with severe heart, kidney, liver or lung failure or other condition that the physician believes may compromise the patient's participation in the study.
* Patient simultaneously participating in another therapeutic trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Continuous Abstinence Rate | Through study completion, an average of 12 months
  Continuous Abstinence Rate within 6 weeks of starting to quit smoking

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France